CLINICAL TRIAL: NCT05838235
Title: Marfan&Moves (M&M's) : an Adapted Physical Activity Program (APA) for Effort Rehabilitation of Children and Teenagers With Marfan Syndrome: an Interventional, Prospective, Monocentric Study.
Brief Title: Adapted Physical Activity Program (APA) for Effort Rehabilitation of Children and Teenagers With Marfan Syndrome
Acronym: M&M's
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RC31/22/0206
Record Dates: First submitted 2023-03-31; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Marfan Syndrome
MeSH Terms: conditions — Marfan Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 6 month adapted physical activity (Experimental): The various assessments will be carried out during 2 visits at 6 months interval as part of the usual follow-up at the Toulouse University Hospital. Standard cardiopulmonary exercise test assessment will be coupled with an assessment by an APA coach on the same day.
  The APA program built from the initial assessment will be returned to the child and his family during a videoconference.
  In addition, a regular reassessment and adjustment of this program will be made every 15 days during phone calls by the APA coach.
  Interventions: Other: Adapted Physical Activity program

INTERVENTIONS:
Other: Adapted Physical Activity program — The Adaptated Physical Activity program will consist of a Personalized Training Program

SUMMARY:
This research study aims to evaluate the effect of a 6-month adapted physical activity program (APA) on the endurance capacities (evaluated as the maximum oxygen consumption [VO2 peak] on a cardiopulmonary exercise test) of children and adolescents with Marfan syndrome or related.

DETAILED DESCRIPTION:
Marfan syndrome (MFS) is characterized by the association of multisystem damage related to connective tissue fragility. The risk of aortic dissection has diverted attention from significant musculoskeletal damage despite commonly reported extreme fatigue and pain with impact on the patient's quality of life. In a recent study (Marfanpower, NCT03236571), investigators have observed reduced endurance capacities in children and teenagers with MFS (average VO2 peak at 60% of expected), which were significantly increased by an intensive rehabilitation program. Based on this experience, investigators aim to evaluate the effect of a physical activity program adapted to the daily life of the young patients on their endurance capacities and their quality of life. This program will be set up by an adapted physical activity (APA) coach after a complete assessment, including a cardiopulmonary exercise test with VO2 peak measurement, which will be carried out in the Reference Centre for Marfan syndrome at the Toulouse University Hospital. The VO2 peak evolution will be evaluated after 6 months of program. This is a recognized parameter for the evaluation of endurance and has been validated in children. Investigators hypothesize that the implementation of a physical activity program adapted to the daily life and interests of the child with MFS will efficiently improve endurance, prevent deconditioning and promote long term benefits.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed Marfan syndrome or related syndrome
* Girl or boy aged 7 to 17
* Informed and written consent signed by at least one of the two holders of parental authority
* Patient affiliated to a social security scheme or equivalent

Exclusion Criteria:

* Cardiac contraindications to the APA program:

  * Severe aortic dilation (aortic diameter > 45 mm)
  * and/or left ventricular failure (left ventricular ejection fraction <45%)
  * and/or severe mitral leakage ≥ grade 3
* Pregnancy

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Measurement of maximum endurance | At baseline
  maximum oxygen consumption (VO2 peak) during a cardiopulmonary exercise test will be measured
Measurement of maximum endurance | Up to 6 month
  maximum oxygen consumption (VO2 peak) during a cardiopulmonary exercise test will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Thomas EDOUARD, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France